CLINICAL TRIAL: NCT02845141
Title: Synthetic Bone Graft Substitute (Actifuse) vs. Autologous Spongiosa for Tunnel Enlargement in Revision Anterior Cruciate Ligament Reconstruction - a Histological and Radiological Assessment
Brief Title: Synthetic Bone Graft Substitute vs. Autologous Spongiosa in Revision Anterior Cruciate Ligament Reconstruction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Berufsgenossenschaftliche Unfallklinik Ludwigshafen (Other)
Responsible Party: Principal Investigator, Jan von Recum, Dr. med., Berufsgenossenschaftliche Unfallklinik Ludwigshafen
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Baxter_Actifuse_001
Record Dates: First submitted 2012-10-13; First posted 2016-07-27 (Estimated); Last update posted 2018-01-19 (Actual); Status verified 2018-01

CONDITIONS: Anterior Cruciate Ligament Injury
Keywords: ACL; Revision surgery; tunnel enlargement; bone substitute material; bone graft
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries | interventions — actifuse synthetic bone graft; Bone Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Actifuse (Experimental): Actifuse to fill bone tunnel
  Interventions: Procedure: Actifuse
- bone graft (Active Comparator): bone graft to fill bone tunnel
  Interventions: Procedure: bone graft

INTERVENTIONS:
Procedure: Actifuse — bone tunnel filled with Actifuse
  Other Names: Baxter Actifuse MIS
  Arms: Actifuse
Procedure: bone graft — bone graft to fill bone tunnel
  Arms: bone graft

SUMMARY:
The overall objective is the histological and radiological assessment of bony consolidation of the tibial/femoral tunnel using either bone graft substitute (Actifuse) or autologous spongiosa in patients undergoing revision anterior cruciate ligament reconstruction.

Clinical correlation with the histological and radiological results using the SF36 questionnaire.

DETAILED DESCRIPTION:
* Study design: Monocentric, prospective, randomised study. Patients who need revision anterior cruciate ligament reconstruction and show a tunnel enlargement of >10mm will have a first operation filling the tibial/femoral tunnel either with bone graft substitute (Actifuse) or autologous spongiosa.

5 - 6 months after this first operation a CT will be performed to assess the bony consolidation of the former tibial/femoral tunnel. An MRI will be performed to assess vitality of the bone substitute.

An osseous biopsy will be taken from the tibial/femoral tunnel at the revision anterior cruciate ligament reconstruction approximately 6 months after bone grafting.

Clinical evaluation will be performed 6 weeks, 3 months and 6 months postoperative. At 6 months postoperative additional radiological evaluation and clinical assessment using the SF36 questionnaire will be performed.

* Treatment: Either autologous spongiosa or Actifuse (MIS applicator) will be administered by the investigator as a bone graft substitute for tunnel enlargement in patients undergoing revision anterior cruciate ligament reconstruction.
* Duration of Participation: The participation of each subject will be approximately 12 months.

Each subject will undergo revision anterior cruciate ligament reconstruction approximately 6 months after bone grafting. A biopsy will be taken at this operation. A clinical and radiological follow up is planned for further 6 months.

* Subjects: Male and female patients ≥ 18 years. Approximately 40 patients who undergo revision anterior cruciate ligament reconstruction will be included in the study.

Inclusion criteria: Patients in need of revision anterior cruciate ligament reconstruction Exclusion criteria: Infection, wound healing complications

ELIGIBILITY:
Inclusion Criteria:

* Patients in need of revision anterior cruciate ligament reconstruction

Exclusion Criteria:

* Infection, wound healing complications

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2013-03; Primary Completion 2016-09 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
histological assessment of bony consolidation | 6 months postop
  histological probes during second intervention to measure bony ingrowth into bone substitute material

SECONDARY OUTCOMES:
Tegner Activity Score | 3, 6 and 12 Months
  functional score
IKDC Score | 3, 6 and 12 Months
  functional score
stability measurement using KT1000 | 3, 6 and 12 Months
  functional score
SF36-Score | 3, 6 and 12 Months
  health score

CONTACTS AND LOCATIONS:
Overall Officials: Jan von Recum, MD, Principal Investigator — BG Unfallklinik Ludwigshafen; Marc Schnetzke, MD, Study Chair — BG Unfallklinik Ludwigshafen
Locations (1):
- BG Unfallklinik, Ludwigshafen, Germany

IPD SHARING:
Plan to Share IPD: No